CLINICAL TRIAL: NCT06349668
Title: SMILe: Spinal Morphine or Intravenous Lidocaine in Robot-assisted Upper Urologic Surgery
Brief Title: Spinal Morphine or Intravenous Lidocaine in Robot-assisted Upper Urologic Surgery
Acronym: SMILe
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hans Bahlmann (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor-Investigator, Hans Bahlmann, Senior Consultant. Sponsor, University Hospital, Linkoeping
Organization: University Hospital, Linkoeping (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-505941-21-00
Record Dates: First submitted 2024-03-24; First posted 2024-04-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Other Specified Disorders of Kidney and Ureter; Benign Neoplasm of Ureter; Calculus of Kidney and Ureter; Ureter Cancer; Ureteric Reflux; Congenital Ureteric Anomaly; Benign Renal Neoplasm; Renal Cancer
MeSH Terms: conditions — Nephrolithiasis; Ureteral Neoplasms; Vesico-Ureteral Reflux; Kidney Neoplasms | interventions — Morphine; Bupivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- spinal analgesia (Experimental): single shot spinal analgesia with 0.2-0.3 mg morphine and 10-20 mg bupivacaine before surgery
  Interventions: Drug: spinal analgesia with morphine and bupivacaine
- lidocaine infusion (Active Comparator): intraoperative intravenous infusion of lidocaine at a rate of 2 mg/kg/t (Ideal Body Weight)
  Interventions: Drug: lidocaine infusion

INTERVENTIONS:
Drug: spinal analgesia with morphine and bupivacaine — single shot spinal analgesia with 0.2-0.3 mg morphine and 10-20 mg bupivacaine before surgery
  Other Names: morphine spinal
  Arms: spinal analgesia
Drug: lidocaine infusion — intraoperative intravenous infusion of lidocaine at a rate of 2 mg/kg/t after a bolus of 2 mg/kg (Ideal Body Weight if BMI > 22, otherwise ABW)
  Other Names: xylocaine iv
  Arms: lidocaine infusion

SUMMARY:
The goal of this clinical trial is to learn whether the addition of spinal analgesia leads to superior recovery in patients undergoing robotic-assisted laparoscopic upper urinary tract surgery under general anesthesia. The main questions it aims to answer are:

* Is the decrease in wellbeing as quantified by the patient-centered outcome scale "Quality of Recovery 15" (QoR-15), from baseline to the first day after surgery (POD 1), at least 8.0 points less in patients receiving spinal analgesia in addition to general anesthesia?
* Does spinal analgesia result in improved recovery as quantified by QoR-15 at POD 7, the incidence of postoperative pain at rest and at mobilization, nausea and vomiting, the need for opioid analgesics, time out-of-bed, length of stay and the incidence of complications?
* Does spinal analgesia increase workload in the OR, as quantified by time from arrival in the OR to start of surgery?
* Does spinal analgesia result in an increased incidence of hypotension and cardiac dysfunction during surgery, as well as an increased incidence of pruritus after surgery?

Participants will be randomized to receive either spinal analgesia with bupivacaine and morphine preoperatively or an intravenous infusion with lidocaine intraoperatively.

QoR-15 and other markers of recovery will be registered using structured interviews preoperatively, at POD1 and POD7. In addition, patients will record pain at rest and at mobilization three times daily in a diary.

In a subgroup of patients advanced hemodynamic parameters will be recorded using pulse-contour analysis before, during and after surgery. Blood samples will also be collected in these patients at fixed intervals and analyzed for amongst others inflammation and cardiac dysfunction.

DETAILED DESCRIPTION:
Please refer to CTIS

ELIGIBILITY:
Inclusion Criteria:

* The patient is scheduled for elective robotic-assisted upper urinary tract surgery at one of the participating hospitals
* The patient gives oral and written informed consent after having received oral and writen information about the study

Exclusion Criteria:

* The patient has a ASA-class of IV or above
* The patient is a minor or declared incompetent, has severe psychiatric disease or is expected not to be able to understand the study information due to severe restrictions in vision, hearing, cognition, reading or Swedish language abilities
* The patient is a female who is pregnant or breastfeeding
* The patient is a pre-menopausal female who has not undergone sterilisation, hysterectomy, bilateral salpingectomy and/or bilateral oophorectomy, and is not using highly-effective contraception with low user-dependency and cannot provide a negative pregnancy test
* The patient is scheduled for emergency surgery
* Research staff not available
* Scheduled significant simultaneous surgery on another organ
* The anesthesiologist in charge has planned spinal or epidural analgesia
* The patient has clear contraindications to spinal analgesia, e.g. severe coagulopathy, severe aortic stenosis, previous back surgery with rods, or spinal analgesia can be expected to be technically challenging (severe obesity, severe scoliosis)
* The patient has clear contraindications to lidocaine infusion, e.g. proven allergy to local anesthetics, myasthenia gravis, renail failure (eGFR < 30), hepatic failure caused by acute hepatitis or cirrhosis (Child-Pugh B or higher, severe cardiac arrythmias or insuffiency (NYHA IIIb or higher)
* The patient has previously participated in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
QoR-15 score at postoperative day 1 | First day after surgery
  Quality of Recovery-15 score ranges from 0 to 150 with 0 reflecting zero wellbeing and 150 reflecting perfect wellbeing. The primary research hypothesis is that the reduction in QoR-15 from baseline before surgery to the first postoperative day (POD 1) is at least 8.0 points less in the morphine spinal group compared to the control group treated with intravenous lidocaine.

SECONDARY OUTCOMES:
QoR-15 score preoperatively | Any time between inclusion and the night before surgery
  Quality of Recovery-15 score ranges from 0 to 150 with 0 reflecting zero wellbeing and 150 reflecting perfect wellbeing.
QoR-15 score at postoperative day 7 | Seventh day after surgery
  Quality of Recovery-15 score ranges from 0 to 150 with 0 reflecting zero wellbeing and 150 reflecting perfect wellbeing.
Pain (NRS) in rest and during motion 2hrs after arrival to the PACU/ICU/HDU | 2 hrs after arrival to the PACU
  Numeric Rating Scale ranges from 0 to 10 with 0 reflecting absence of pain and 10 reflecting extreme pain.
Pain (NRS) on POD 1-3 | First, second and third day after surgery
  Numeric Rating Scale ranges from 0 to 10 with 0 reflecting absence of pain and 10 reflecting extreme pain.
Pain (NRS) in rest and during motion at POD 7 | Seventh day after surgery
  Numeric Rating Scale ranges from 0 to 10 with 0 reflecting absence of pain and 10 reflecting extreme pain.
Time from arrival in the OR to start of surgery | Time from entering the OR to first incision or start of endoscopy, whichever comes first, up to 4 hrs.
  Time from entering the OR to first incision or start of endoscopy, whichever comes first, up to 4 hrs.
Time from end of surgery until leaving the OR | Time from end of surgery (removing of surgical drapes or finishing of endoscopy, whichever comes last) until leaving the OR, up to 4 hrs
  Time from end of surgery (removing of surgical drapes or finishing of endoscopy, whichever comes last) until leaving the OR, up to 4 hrs
Incidence of unplanned termination of the lidocaine infusion | Intraoperatively
  Incidence of unplanned termination of the lidocaine infusion
Amount of remifentanil in patients given remifentanil | Intraoperatively
  Amount of remifentanil during anesthesia in patients given remifentanil expressed in mcg/kg/min as recorded on the anesthetic chart.
Amount of intraoperative opioids in patients not receiving remifentanil | Intraoperatively
  Amount of intraoperative opioids in patients not receiving remifentanil expressed in mcg/kg/min morphine equivalents as recorded on the anesthetic chart.
Length of stay at the PACU/ICU/HDU | Length of stay at the PACU (from first to final recording of any vital sign by the electronic patient data management system), up to 30 days
  Length of stay at the PACU/ICU/HDU (from first to final recording of any vital sign by the electronic patient data management system), up to 30 days
Amount of opioids administred at the PACU/ICU/HDU during the first 24 hrs after end of surgery | During stay at the PACU (from first to final recording of any vital sign by the electronic patient data management system), up to 30 days
  Amount of opioids administered at the PACU/ICU/HDU expressed in mcg/kg morphine equivalents as recorded on the post-anesthetic chart.
PONV requiring treatment at 0-6 hours and 6-24 hours postoperatively as well as during the whole postoperative stay | At 0-6 hours and 6-24 hours postoperatively as well as during the whole postoperative stay
  PONV requiring treatment at 0-6 hours and 6-24 hours
"Time out-of-bed" on POD 1-3 | First, second and third day after surgery
  "Time out-of-bed" on POD 1-3
Amount of opioids administered during the first 24 hours at the PACU/ICU/HD and on the ward | During the first 24 hours at the PACU and on the ward
  Amount of opioids expressed in mcg/kg morphine equivalents administered during the first 24 hours at the PACU/ICU/HD and on the ward as recorded on the ward chart.
First POD passing gases | From first until seventh day after surgery
  First POD passing gases
First POD passing stool | From first until seventh day after surgery
  First POD passing stool
Incidence of pruritus | From first until seventh day after surgery
  Incidence of pruritus
Length of stay | From first until thirtieth day after surgery
  Length of stay in calendary days
DAOH30 | From first until thirtieth day after surgery
  Days Alive and Out of Hospital defined as the number of full calendary days where the patient is not admitted to a hospital and not deceased
Postoperative complications untill POD 30 | From first until thirtieth day after surgery
  Postoperative complications untill POD 30
Requirement for opioids after discharge | From first until seventh day after surgery
  Y/N, based on a telephone interview
Incidence of respiratory depression leading to the use of a mu-antagonist within 48 hours of induction of anesthesia | From induction of anesthesia until 48 hours after induction of anesthesia
  Incidence of respiratory depression leading to the use of a mu-antagonist within 48 hours
Intraoperative fluid balance | Intraoperatively
  Intraoperative fluid balance as recorded on the CRF in ml, defined by the estimated sum of administered fluids minus estimated bleeding, diuresis and other measurable losses.
Time with low blood pressure during anesthesia | Intraoperatively
  Time with low blood pressure during anesthesia
Lowest MAP within 10 minutes after induction of anesthesia | Within 10 minutes after induction of anesthesia
  Lowest MAP within 10 minutes after induction of anesthesia
Highest MAP within 10 minutes of start of abdominal insufflation | Within 10 minutes of abdominal insufflation
  Highest MAP within 10 minutes of start of abdominal insufflation
Fraction of patients needing norepinephrine within 15 minutes after start of abdominal insufflation | From anesthesia induction until 15 minutes after start of abdominal insufflation
  Fraction of patients needing norepinephrine within 15 minutes after start of abdominal insufflation
Fraction of patients needing norepinephrine intraoperatively (later than 15 minutes after start of abdominal insufflation) | Intraoperatively (later than 15 minutes after start of abdominal insufflation)
  Fraction of patients needing norepinephrine intraoperatively (later than 15 minutes after start of abdominal insufflation)
Average infusion rate of norepinephrine, in patients receiving norepinephrine, before 15 minutes after start of abdominal insufflation | From anesthesia induction until 15 minutes after start of abdominal insufflation until end of anesthesiaon, up to 48 hours
  Average infusion rate of norepinephrine, in patients receiving norepinephrine, before 15 minutes after start of abdominal insufflation
Average infusion rate of norepinephrine, in patients receiving norepinephrine, after 15 minutes after start of abdominal insufflation | From 15 minutes after start of abdominal insufflation until end of anesthesia (extubation), up to 48 hrs
  Average infusion rate of norepinephrine, in patients receiving norepinephrine, after 15 minutes after start of abdominal insufflation
Intraoperative Cardiac Index | Intraoperative
  Cardiac output corrected for Body Surface Area expressed in L/min/m2
Intraoperative Stroke Volume Index | Intraoperative
  Stroke volume corrected for Body Surface Area expressed in mL/m2
Intraoperative Cardiac Power Index | Intraoperative
  Cardiac Power Output corrected för Body Surface Area, expressed in Watt/m2, with higher values implying better cardiac performance.
Intraoperative dPmx | Intraoperative
  Maximum increase in arterial pressure during a cardiac cycle, expressed in mmHg/second, with higher values implying better cardiac contractility.
Intraoperative Pulse Pressure Variation | Intraoperative
  Determined as the ratio of the difference between the maximal and minimal values of pulse pressure over the mean of these two values and expressed as a percentage
Intraoperative Stroke Volume Variation | Intraoperative
  Determined as the ratio of the difference between the maximal and minimal values of stroke volume over the mean of these two values and expressed as a percentage
Intraoperative dynamic arterial elastance | Intraoperative
  Determined as Pulse Pressure Variation divided by Stroke Volume Variation
Intraoperative Systemic Vascular Resistance Index | Intraoperative
  Intraoperative Systemic Vascular Resistance corrected for Body Surface Area
Intraoperative heart rate | Intraoperative
  Intraoperative heart rate
Biochemical markers of inflammation | Day of surgery and first and third day after surgery.
  To be specified later during the study (samples are stored for later analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Holmberg, Principal Investigator — University Hospital, Linkoeping
Locations (3):
- Sweden (3):
  - Länssjukhuset i Kalmar, Kalmar
  - University Hospital Linköping, Linköping
  - Centrallasarettet Växjö, Vaxjo

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available on reasonable request
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within 2 months of publication of the data involved
Access Criteria: reasonable request